CLINICAL TRIAL: NCT01113424
Title: Bioequivalence Between Oral Nicotine Replacement Products and Nicorette® Gum - A Study in Healthy Smokers
Brief Title: Bioequivalence Between Nicotine Replacement Products and Nicorette® Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP1071; 2008-003358-14 (EudraCT Number)
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NRT-2 (Experimental): 2 mg single-dose of a new NRT product
  Interventions: Drug: Nicotine
- GUM-2 (Active Comparator): 2 mg single-dose of a marketed nicotine gum
  Interventions: Drug: Nicorette® (Nicotine Gum)
- NRT-4 (Experimental): 4 mg single-dose of a new NRT product
  Interventions: Drug: Nicotine
- GUM-4 (Active Comparator): 4 mg single-dose of marketed nicotine gum
  Interventions: Drug: Nicorette® (Nicotine Gum)

INTERVENTIONS:
Drug: Nicotine — Single-dose of a new Nicotine Replacement Therapy (NRT) product 2 mg and 4 mg
  Other Names: Not yet marketed
  Arms: NRT-2; NRT-4
Drug: Nicorette® (Nicotine Gum) — Single-dose of marketed nicotine gum 2 mg or 4 mg
  Other Names: Nicorette®
  Arms: GUM-2; GUM-4

SUMMARY:
Bioequivalence between oral nicotine replacement products and Nicorette® gum.

DETAILED DESCRIPTION:
This study compares a new oral Nicotine Replacement Therapy (NRT) product containing 2 and 4 mg nicotine with Nicorette® gum 2 mg and 4 mg, after 12 hours of nicotine abstinence, with respect to nicotine pharmacokinetics, during 10 hours after start of administration. Single doses of each treatment are given once in the morning during four separate treatment visits scheduled in a crossover setting with randomized treatment sequences. The study will include 88 healthy smokers between 18-50 years, who have been smoking at least 10 cigarettes daily during at least one year preceding inclusion. Subjects and study personnel will be aware of which treatment is administered at a given visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers, smoking at least 10 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurements | Baseline and during 10 hours after product administration
  Pharmacokinetic measurements including:
  * the maximum observed nicotine concentration in plasma (Cmax)
  * the area under the plasma concentration-vs.-time curve until the last measurable concentration (AUCt)
  * the area under the plasma concentration-vs.-time curve until infinity (AUCinf)

SECONDARY OUTCOMES:
Tmax | during 10 hours after start of product administration
  The time of occurrence of Cmax (tmax) following product administration
λz | during 10 hours after start of product administration
  The terminal nicotine elimination rate constant (λz)
Residual Nicotine | After 30 minutes of chewing
  The amount of nicotine released from Nicorette® gum 2 and 4 mg during 30 minutes' chewing.
Dissolution Time | From product administration until completely dissolved
  Actual time required for oral dissolution of new NRT products following product administration

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Berzelius Clinical Research Center, Linköping, Sweden